CLINICAL TRIAL: NCT02037269
Title: A Pilot Study to Evaluate Cerenkov Luminescence Imaging for Measuring Margin and Lymph Node Status in Breast Cancer Surgical Specimens
Brief Title: LightPathTM Imaging System for Ex-vivo Assessment of Margin and Lymph Node Status in Breast Cancer Surgical Specimens
Status: Completed | Type: Observational
Sponsor: Lightpoint Medical Limited (Industry)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: LPM-001
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Cerenkov Luminescence Imaging, CLI, margin status
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Female patients ≥30 years of age with known breast cancer scheduled for breast-conserving surgery (BCS) +/- sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND)

SUMMARY:
This study is a prospective, cross-sectional observational single centre study to assess the feasibility of intra-operative Cerenkov Luminescence Imaging (CLI) of breast cancer wide local excision (WLE) specimens and dissected lymph nodes. The samples will be imaged using the LightPathTM Imaging System. The LightPathTM Imaging System which consists of a light-tight box on which are mounted an ultra-sensitive lens and radiation-shielded camera. This study will measure the correlation between margin status of the WLE specimen and the metastatic status of dissected lymph nodes as determined by the LightPathTM Imaging System and by histopathology. This is a pilot study to assess feasibility before proceeding to a pivotal study to evaluate the benefits of the LightPathTM Imaging System in clinical practice.

DETAILED DESCRIPTION:
Subject's blood glucose level will be measured on the day of surgery. Subjects with a blood glucose level < 12 mmol/l receive an intravenous injection of 5 MBq/kg, up to a maximum 300 MBq of 18F-fluorodeoxyglucose (18F-FDG) prior to surgery. Breast cancer surgery will be performed per standard of care. SLNB will be performed using a dose of 150 MBq technetium 99 (99mTc) nanocolloid and patent blue dye. The resected WLE specimen and lymph nodes will be imaged in the LightPathTM Imaging System. A member of the research team who is not the operating surgeon will capture LightPathTM images intra-operatively.

Prior to CLI, the WLE specimen will be placed in a specimen holder. CLI is performed according to the LightPathTM Imaging System instructions for use. All CLI will be performed between 1 and 3 hours post injection of 18F-FDG.

The WLE specimen will then undergo standard of care histopathological analysis with a positive margin defined as either invasive carcinoma or ductal carcinoma in situ (DCIS) within 2mm of the specimen surface. Lymph nodes will also be examined according to standard of care histopathological analysis.

The CLI results will not be used to influence any surgical or clinical decision-making.

All staff in the operating theatre and the recovery area caring for the patient, and pathology staff processing surgical specimens will wear badge dosimeters. Staff handling surgical specimens will also wear ring dosimeters.

ELIGIBILITY:
Inclusion Criteria

* Females ≥30 years of age with a diagnosis of invasive breast cancer or DCIS
* Scheduled for BCS +/- SLNB or ALND
* Females of childbearing age must have a negative pregnancy test (by Beta HCG qualitative analysis), must have had a history of a surgical sterilisation, or must give history of no menses in past twelve months

Exclusion Criteria

* Surgery or radiotherapy in the operated breast in the past 2 years
* Neoadjuvant systemic therapy
* Patients not suitable for BCS
* Blood glucose level ≥ 12 mmol/l on the day of surgery
* Known hypersensitivity to 18F-FDG
* Any patient who is pregnant or lactating

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients ≥30 years of age with known breast cancer scheduled for breast-conserving surgery (BCS) +/- sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Tumour margin status of the Wide Local Excision specimen as determined by the LightPathTM Imaging System | Intra-operative

SECONDARY OUTCOMES:
Metastatic status of dissected lymph nodes as determined by the LightPathTM Imaging System | Intra-operative
Radiation dosimetry to operating theatre, recovery area and pathology staff | Up to 24 hours after injection of radiopharmaceutical
Ease of use of the LightPathTM Imaging System | Intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Anand D Purushotham, MBBS FRCS MD, Principal Investigator — King's College London
Locations (1):
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grootendorst MR, Cariati M, Pinder SE, Kothari A, Douek M, Kovacs T, Hamed H, Pawa A, Nimmo F, Owen J, Ramalingam V, Sethi S, Mistry S, Vyas K, Tuch DS, Britten A, Van Hemelrijck M, Cook GJ, Sibley-Allen C, Allen S, Purushotham A. Intraoperative Assessment of Tumor Resection Margins in Breast-Conserving Surgery Using 18F-FDG Cerenkov Luminescence Imaging: A First-in-Human Feasibility Study. J Nucl Med. 2017 Jun;58(6):891-898. doi: 10.2967/jnumed.116.181032. Epub 2016 Dec 8. PMID 27932562
- See also: Sponsor website — http://www.lightpointmedical.com/
- See also: Study site web page — http://www.guysandstthomas.nhs.uk/